CLINICAL TRIAL: NCT06861725
Title: CARIES ARREST USING SILVER DIAMINE FLUORIDE VERSUS FISSURE SEALANT in OCCLUSAL DENTAL CARIOUS LESIONS: RANDOMIZED CONTROLLED TRIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Abir Atmaz Alsibaee, Dr.Amr Abir Atmaz Alsibaee, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDF VS FS in caries arrest
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Caries Arrested; Silver Diamine Fluoride; Fissure Sealant
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Masking Description: Biostatistics: The study was divided into two groups, Group A and Group B. The materials used in each group were blinded to the statisticians conducting the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VOCO Fissurit (Active Comparator): Sealants are restorative dental materials applied to the pit-and-fissure surfaces of teeth. Upon application, the sealant material infiltrates the pits and fissures, subsequently polymerizing to form a hardened layer. This layer serves as a physical barrier, effectively preventing or restricting the penetration of bacteria and nutrients, thereby mitigating the risk of caries formation in these susceptible areas. Pit and fissure sealants: Evidence-based recommendations support the use of sealants for the prevention and management of pit and fissure caries. Sealants are effective and should be applied to the occlusal surfaces of first and second permanent molars. Additionally, non-operative cleaning of fissures with a toothbrush or bristle brush is recommended.
  Interventions: Other: VOCO Fissurit
- Silver Diamine Fluoride (SDF) (Experimental): Advantage Arrest Silver Diamine Fluoride 38%-SDF is an anti-microbial and remineralizing liquid clinically applied to control and arrest active dental caries and stop hypersensitivity. It is a safe, painless alternative to traditional cavity drilling procedures with the Power of Silver and Fluoride. Silver acts as an antimicrobial agent that simultaneously strengthens the dentin. Fluoride is the active ingredient that puts a stop to tooth decay by remineralising and helps prevent additional decay from appearing. It is also helpful to get relief from hypersensitivity.
  The only common side effect is SDF causes black staining, but SDF/KI and NSF may reduce this staining effect. SDF can also stain surfaces that it comes into contact with when being applied, such as clothing or nearby tissues in the mouth. For best results, SDF should be reapplied every 3, 6, or 12 months, If the cavity still progresses.
  Interventions: Other: Silver Diamine Fluoride (SDF)

INTERVENTIONS:
Other: Silver Diamine Fluoride (SDF) — Silver Diamine Fluoride has been used extensively around the globe for decades. Advantage Arrest silver diamine fluoride 38% will change how you offer your patients the protection they deserve.
  Advantage Arrest:
  Provides immediate relief from dentinal hypersensitivity Kills pathogenic organisms Hardens softened dentin making it more acid and abrasion resistant Does not stain sound dentin or enamel Can provide important clinical feedback due to its potential to stain visible or hidden lesions Silver diamine fluoride 38% is indicated for the treatment of dentinal hypersensitivity.
  Arms: Silver Diamine Fluoride (SDF)
Other: VOCO Fissurit — Transparent Light-cured pits and fissure sealant, with high stability and good adhesion to enamel
  Arms: VOCO Fissurit

SUMMARY:
The goal of this randomized clinical trial is to evaluate if Silver Diamine Fluoride (SDF) is a more conservative and effective treatment in preventing the progression of mild occlusal caries compared to fissure sealant in patients aged 20-45 years with incipient molar caries. The main question it aims to answer is:

Is SDF more effective in arresting caries progression than fissure sealant? Does SDF prevent the formation of new caries compared to fissure sealant? Researchers will compare SDF treatment to fissure sealant application to see if SDF results in better caries arrest and fewer new carious lesions.

Participants will:

Be randomly assigned to receive either SDF or fissure sealant. Have follow-up assessments at 1, 3, 6, and 12 months for caries progression, arrest, and new caries formation.

Undergo clinical evaluations using visual and tactile examinations to assess caries arrest and progression and using DIAGNOdent laser fluorescence system .

DETAILED DESCRIPTION:
This randomized clinical trial aims to assess the efficacy of Silver Diamine Fluoride (SDF) compared to fissure sealant in arresting mild occlusal caries. The study is focused on patients aged 20 to 45 years who present with incipient caries in the molar teeth, classified under ICDAS 1 and 2. The study will be conducted at the Cairo University Dental Hospital, a tertiary healthcare and referral center.

The null hypothesis is there is no difference in the clinical performance between the application of silver diamine fluoride and fissure sealant in occlusal dental carious lesions.

Participants will be randomly assigned to one of two groups:

SDF Group: Silver Diamine Fluoride (38%) will be applied to the affected tooth surface. The treatment will be carried out by isolating the tooth, drying it thoroughly, applying SDF using a microbrush, and allowing it to remain on the surface for up to 3 minutes. Afterward, any excess will be removed, and the patient will be advised to avoid eating for 30 minutes.

Fissure Sealant Group: Fissure sealant (resin-based) will be applied to the affected occlusal surface. This procedure involves etching the surface with phosphoric acid, applying the sealant, and then curing it using a light-curing device. The sealant will form a protective barrier to prevent further demineralization.

The study will track two primary outcomes:

Caries progression, measured by the presence of visible cavitation or sensitivity during follow-up.

Caries arrest, determined through visual and tactile examination (e.g., probing to assess lesion hardness).

Secondary outcomes will include the formation of new caries, assessed using the DIAGNOdent laser fluorescence system.

Follow-up visits will occur at 1, 3, 6, and 12 months, where participants will be clinically assessed for pain, caries arrest, and new lesions. Clinical evaluations will include:

Visual and tactile examinations: Assessing the presence and activity level of carious lesions.

Caries progression: Identified by tactile detection with a dental explorer. Caries arrest: Lesions that have become hard and smooth will be considered arrested.

New caries: Monitored using the DIAGNOdent system for any signs of new decay. This trial will provide insight into whether SDF, a minimally invasive treatment, can offer a more effective and less expensive alternative to fissure sealants in arresting caries, especially in patients with early-stage occlusal caries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consulting in the outpatient clinic.
2. Patients with enamel caries in molars permanent teeth, according to ICDAS 1 and 2.
3. Provide informed consent.
4. Co-operative patients approving to participate in the trial.
5. Patient age (20-45 years old).

Exclusion Criteria:

1. Tooth mobility.
2. Signs of pulpal infection.
3. Severe medical conditions that would not allow management in the clinic.
4. Hereditary developmental defects, such as amelogenesis imperfecta or dentinogenesis imperfecta.
5. Known allergies or sensitivities to dental materials, including SDF and fissure sealant.
6. Inability to return for recall visits.
7. Patients with bad oral hygiene
8. Refuse to participate in the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
detect clinical progression done by the presence of visible cavitation and/or sensitivity during follow-up, measured by visual criteria | 1-3-6 and 12 month
  detect clinical progression done by the presence of visible cavitation and/or sensitivity during follow-up, measured by visual criteria.
  The fissure sealant and SDF will be evaluated at each recall visit for caries arrest through visual and tactile assessment, Arrested caries treated with silver diamine fluoride is clinically characterized by increased hardness and dark brown to black coloration . The clinical examination of fissure sealants involved evaluating the presence of visible cavitation. Although lesions can be seen through sealants.
  Active caries will be identified when a blunt probe, applied with light pressure, can easily penetrate the lesion surface. Conversely, inactive (arrested) caries will be observed if the lesion surface is firm, smooth, and free from plaque. The number and percentage of arrested carious lesions will be recorded and assessed.

SECONDARY OUTCOMES:
evaluate carries arrest and new caries formation, measured by DIAGNOdent laser fluorescence system | 1-3-6 and 12 month
  The DIAGNOdent system provides fluorescence scores that range from 0 to 99. These scores indicate the level of caries activity or demineralization in the tooth structure.
  -Score 0-13: Healthy Tooth Structure
  -Score 14-20: Early Demineralization/Initial Lesion Mild demineralization is present, which may be reversible. These lesions might not be cavitated but show early signs of enamel breakdown..
  -Score 21-40: Moderate Demineralization Clear signs of enamel breakdown, but the lesion is still confined to the enamel without progressing to the dentin.
  -Score 41-60: Active Lesion Significant demineralization is occurring.
  -Score 61-99: Cavitation and Severe Active Caries Indicates severe decay or active caries.

CONTACTS AND LOCATIONS:
Overall Officials: Omaima Safwat Hamza, Professor, Study Director — Professor of Esthetic and Conservative Dentistry, Faculty of Dentistry, Cairo University in Egypt.; Dina Mounir El-Kadi, Study Director — Lecturer of Esthetic and Conservative Dentistry, Faculty of Dentistry, Cairo University.

IPD SHARING:
Plan to Share IPD: Yes